CLINICAL TRIAL: NCT03191877
Title: Effect of Coffee Consumption on Intestinal Motility After Caesarean Sections; Randomized Controlled Trial
Brief Title: Effect of Coffee Consumption on Intestinal Motility
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Armed Forces Hospitals, Southern Region, Saudi Arabia (Other Government)
Responsible Party: Principal Investigator, Mufareh Asiri, OB/GYN REGISTRAR, Armed Forces Hospitals, Southern Region, Saudi Arabia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: H-06-KM-001
Record Dates: First submitted 2017-06-09; First posted 2017-06-19 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2017-06

CONDITIONS: Gastrointestinal Motility
Keywords: coffee consumption; Cesarean section; intestinal motility
MeSH Terms: interventions — Coffee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- COFFEE (Experimental): they will start to drink coffee 6 hours postoperative for maximum 3 doses (100ml), 8 hours apart, diet will start after 1st audible bowel sound.
  Interventions: Dietary Supplement: coffee
- oral fluid (Active Comparator): they will drink plain fluid (water) 6 hours postoperative. Diet will start after 1st audible bowel sound.
  Women in this group will not receive either coffee.
  Interventions: Dietary Supplement: coffee
- control (No Intervention): the control group and they will be NPO for 24 hours on IV fluid (3 LITRES/24 HOURS). Diet will start after 1st audible bowel sound

INTERVENTIONS:
Dietary Supplement: coffee — Nescafe "brand of coffee made by Nestlé", red mug 100 % pure coffee 12083811
  Arms: COFFEE; oral fluid

SUMMARY:
Randomized controlled trial in Obstetrics and Gynecology department (MULTI-CENTRIC).To measure the effect of coffee consumption on intestinal motility after caesarean section for the patient who fulfills the criteria. Then they will be randomized to 3 groups. The primary outcome and secondary outcome will be measured.

DETAILED DESCRIPTION:
Randomized controlled trial. Participants who fulfill the inclusion criteria (elective caesarian section, singleton pregnancy, term, viable fetus), and exclusion criteria (medical disorders, known intestinal diseases, past history of intestinal surgery, intraoperative diagnosis of extensive adhesion, intraoperative complications "e.g., intestinal injury and ureteric injury intraoperative complication that can lengthen the operation time, postoperative complications like anesthesia complication and electrolytes imbalance ) Then they will be randomized to 3 groups. Group 1, will start to drink coffee 6 hours postoperative for maximum 3 doses (100ml), 8 hours apart, diet will start after 1st audible bowel sound.

Group 2, will drink water 6 hours postoperative. Diet will start after 1st audible bowel sound.

Group 3 is the control group and they will be (NOTHING PER ORAL) for 24 hours on intravenous fluid (3 LITRES/24 HOURS). Diet will start after 1st audible bowel sound.

Primary outcome: passage of stool. Secondary outcome: passage of flatus, audible intestinal sound time, feeding time, pain scale by Visual Analogue Scale (VAS), amount, and type of analgesia needed, breastfeeding time, mobilization and hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* elective caesarian section, singleton pregnancy, term, viable fetus

Exclusion Criteria:

* medical disorders, known intestinal diseases, past history of intestinal surgery, intraoperative diagnosis of extensive adhesion, intraoperative complications "e.g., intestinal injury and ureteric injury intraoperative complication that can lengthen the operation time, postoperative complications like anesthesia complication and electrolytes imbalance )

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2018-01-09 (Estimated); Primary Completion 2018-05-30 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
passage of stool. | 72 hours
  passage of stool within 72 hours. (time to be recorded by 24-hour clock from finishing of surgery)

SECONDARY OUTCOMES:
Passage of flatus. . The amount of analgesia. The first Breastfeeding time. The initiation of Mobilization. Hospital length stay. | 72 hours
  (time to be recorded by the 24-hour clock from finishing of surgery).
Audible intestinal sound time. | 72 hours
  Audible first intestinal sound time.(time to be recorded by the 24-hour clock from finishing of surgery).
Feeding time | 72 hours
  Feeding time (StARTING OF REGULAR DIET ).(time to be recorded by the 24-hour clock from finishing of surgery).
Pain scale by VAS (Visual Analogue Scale ). | 72 hours
  Pain scale by using Visual Analogue Scale(VAS). it is measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100.
  No pain (0-4 mm), mild pain (5-44 mm), moderate pain (45-74 mm), and severe pain (75- 100 mm).
Type of analgesia needed. | 72 hours
  Type of analgesia needed. (paracetamol, nonsteroidal anti-inflammatory drugs or pethidine ).
The amount of analgesia . | 72 hours
  ( recording of dose and frequency in time are mandatory ).
The first Breastfeeding time. | 72 hours
  (time to be recorded by 24-hour clock from finishing of surgery)
The initiation of Mobilization. | 72 hours
  (time to be recorded by 24-hour clock from finishing of surgery)
Hospital length stay. | 72 hours
  ( in Days )

CONTACTS AND LOCATIONS:
Overall Officials: Mufareh Asiri, SBOG, Study Chair — Postpartum ward of Armed Forces Hospital, Southern Region. Khamis Mushait, Asir, Saudi Arabia, 101
Locations (1):
- AFHSR, Khamis Mushait, Abha, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided